CLINICAL TRIAL: NCT06671899
Title: Nineteen Years of Modified Constraint-Induced Movement Therapy in a Clinical Setting
Brief Title: Nineteen Years of Modified CIMT in a Clinical Setting, to Improve Arm and Hand Function After Stroke
Status: Completed | Type: Observational
Sponsor: Region Jönköping County (Other Government)
Collaborators: Futurum - Academy for health and care (Unknown)
Responsible Party: Principal Investigator, Maria Landén, Registered Physiotherapist, Master of Science, Region Jönköping County
Other Study IDs: 2019-02250
Record Dates: First submitted 2024-10-15; First posted 2024-11-04 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Neurological Diseases or Conditions
Keywords: stroke rehabilitation; physiotherapy; occupational therapy; neurological rehabilitation; upper extremity; CIMT; CI therapy
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIMT in a clinical setting: Those who underwent modified constraint-induced movement therapy in a clinical setting in Sweden during the years 2000-2018.
  Interventions: Other: Constraint-induced movement therapy (CIMT)

INTERVENTIONS:
Other: Constraint-induced movement therapy (CIMT) — Clinically implemented modified CIMT. Including the three main components; intensive and repetitive task-oriented training of the affected limb, constraint of the non-affected limb and behavioural strategies known as the Transfer Package. In this model the training is supervised by therapist from several professions and some training sessions is performed in group settings with other inpatients and outpatients undergoing primary rehabilitation at the clinic.

SUMMARY:
The goal of this observational study is to determine if clinically constraint-induced movement therapy (CIMT), when applied in a routine clinical practice, can improve arm- and hand function after stroke. Additionally, the study seeks to identify which patients experienced the greatest improvements, and to examine factors that contribute to the long-term sustainability of the treatment.

Stroke is one leading cause of disability, often resulting in difficulties using the arm and hand function on one side, making daily activities challenging. CIMT aims to enhance arm and hand function after stroke by incorporating intensive training and restraining the non-affected limb, thereby encouraging the use of the affected arm and hand. While numerous studies have demonstrated the effectiveness of CIMT, and it is recommended in national clinical guidelines, it is rarely implemented in clinical practice due to challenges in execution and sustainability. Moreover, it remains unclear which patients benefit the most from the treatment.

At a rehabilitation clinic in Sweden, CIMT has been incorporated into routine care for 19 years, which is uncommon. Participants undergo CIMT as outpatients over a three-week period, with one patient being treated at a time. By retrospectively observe outcomes from this clinically implemented and sustained model of CIMT, the study aims to address the following questions:

* Is CIMT, when conducted in a regular clinical setting, effective?
* Are there relationships between patient characteristics and outcomes?

ELIGIBILITY:
Inclusion Criteria:

* Post-acute injury (participants had completed primary rehabilitation and were living at home)
* Reduced ability to use the hemi-paretic arm
* Ability to actively extend the metacarpophalangeal and the interphalangeal joints 10°
* Ability to actively extend the wrist 20°

Exclusion Criteria:

* Unable to walk and balance safely without using the non-affected hand, with or without a mobility aid
* Unable to understand the content of the training or lack of motivation
* Serious cognitive deficit or instable medical condition believed to affect training participation
* Pain in the affected arm believed to affect training intensity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing upper extremity impairments following neurological disorders who underwent a CIMT program at a multidisciplinary rehabilitation medicine clinic in Jönköping, Sweden during the years 2000 and 2018.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2000-08-14 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
The Patient-Specific Functional Scale (PSFS) | From start to the end of treatment at 3 weeks, and at follow-up at 6 months.
  The Patient-Specific Functional Scale is a self-reporting tool meticulously designed to capture and document activity performance challenges identified as significant by the patient. The patients rate their performance on a numeric rating scale from 0 to 10 (0, unable to perform activity; 10, able to perform activity without difficulties or at pre-injury level). In this study, patients autonomously selected 1-5 activities aligned with their personal goals and rated their performance using the PSFS (a mean score for the self-identified activities was labelled PSFS-self). Additionally, patients assessed a single predetermined activity, namely eating with a knife and fork; which was included in the exercise programme for all patients on a daily basis (labelled PSFS-KF).

SECONDARY OUTCOMES:
Motor Activity Log (MAL) | From start to the end of treatment at 3 weeks, and at follow-up at 6 months.
  MAL evaluates daily hand use. MAL consists of two assessment subscales including 30 common daily tasks (0, no use of the affected extremity; 5, normal use). The results are presented as mean values. One subscale concerns the quality of movement (QOM) and one subscale concerns the amount of use. In this study, only the MAL QOM subscale was applied.
The Box and Block Test (BBT) | From start to the end of treatment at 3 weeks, and at follow-up at 6 months.
  The Box and Block Test (BBT) was used to measure gross manual dexterity. The test consists of a box with two compartments and 150 small blocks. The patient grasps and transport the blocks from one compartment to the other. The test score is the number of blocks transported in 60 s.
BL motor assessment | From start to the end of treatment at 3 weeks, and at follow-up at 6 months.
  BL motor assessment is a measurement of motor function after stroke, modified after the Fugl-Meyer Assessment Scale. It includes assessment of the ability to perform active movements and rapid movement changes, balance, sensation, mobility, joint pain and passive range of motion. The test includes several parts but only the upper extremity active movements subpart for the affected side (maximum score 57 points) was used in this study. Each item score from 0 (no ability) to 3 (normal function) and the sum score is used with a maximum score for each side of 57 points for an upper extremity.
Active range of motion (AROM) | From start to the end of treatment at 3 weeks, and at follow-up at 6 months.
  Active range of motion (AROM) was measured using a conventional goniometric technique (Hoppenfeld & Hutton, 1976). The following joint movements were selected because of their big impact on daily activities: shoulder flexion, shoulder abduction, shoulder external rotation, elbow extension, supination and wrist extension. With no compensatory movements allowed, in a sitting position, the maximum AROM was measured and recorded in degrees.
Modified Ashworth Scale (MAS) | From start to the end of treatment at 3 weeks, and at follow-up at 6 months.
  Spasticity in elbow and wrist flexors was assessed with the 6-level modified Ashworth Scale. The therapist measures the resistance to passive movement of a relaxed group of muscles and characterizes change in muscle tone (0, no increase in spasticity; 5, affected part is rigid in flexion or extension).

CONTACTS AND LOCATIONS:
Overall Officials: Kersti Samuelsson, Assoc.Prof., Study Chair — Department of Health, Medicine and Caring Sciences, Linköping University, Linköping, Sweden
Locations (1):
- Department of Rehabilitation Medicine, Region Jönköping County, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: No